CLINICAL TRIAL: NCT06433076
Title: The Association Between Respiratory Effort Parameters During the First 48 Hours With Clinical Outcomes in Mechanically Ventilated Patients: A Prospective Observational Study.
Acronym: EFFORT-1
Status: Completed | Type: Observational
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Phruet Soipetkasem, Critical care medicine, Ramathibodi Hospital
Other Study IDs: COA. MURA2022/317
Record Dates: First submitted 2024-05-19; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Effort; Respiratory Distress Syndrome; Lung Mechanics
Keywords: Respiratory effort; Acute respiratory distress syndrome (ARDS); Dynamic transpulmonary pressure swing (Predicted ΔPL); Patient self-inflicted lung injury (P-SILI); Patient ventilator asynchrony (PVA)
MeSH Terms: conditions — Respiratory Distress Syndrome; Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preference respiratory effort: The preference respiratory effort group was defined by either 1.5≤P0.1≤3.5 cmH2O, 5≤ predicted Pmus≤10 cmH2O, or predicted ΔPL≤20 cmH2O.
- Insufficiency respiratory effort: The insufficiency respiratory effort group was defined by either P0.1<1.5 cmH2O or predicted Pmus < 5 cmH2O.
- Excessive respiratory effort: The excessive respiratory effort group was defined by either P0.1 > 3.5 cmH2O, predicted Pmus > 10 cmH2O, or predicted ΔPL > 20 cmH2O.

SUMMARY:
Over-assisted mechanical ventilation (MV) is linked to respiratory muscle disuse atrophy, while under-assisted MV can lead to patient self-inflicted lung injury (P-SILI) or respiratory muscle injuries. Both scenarios result in poor outcomes. This hypothesis aims to demonstrate the association between the degree of respiratory effort which was measured by P0.1, predicted Pmus, and predicted Δtranspulmonary pressure (ΔPL) with ventilator-free days (VFD) and 28-day mortality.

DETAILED DESCRIPTION:
Recently, the lung and diaphragm protective strategy is an important consideration when providing mechanical ventilation to critically ill patients. Although mechanical ventilation can be life-saving, improper management can cause harm. The harmful mechanical ventilator setting can result from over-assisted or under-assisted ventilation. Over-assisted ventilation can be caused by too much ventilatory support or calming down patients with high dosages of sedative drugs or muscle relaxants, which negatively affect the operation of the diaphragm leading to diaphragm muscle atrophy and weakness. This can make it more difficult to weaning and lead to prolonged use of mechanical ventilation. It appears that previous study found a correlation between percentage change in diaphragm thickness fraction, as measured by ultrasound, during the first week of mechanical ventilation and prolonged duration of mechanical ventilation, extended length of stay in the ICU, and complications. Additionally, in the study conclusions, a diaphragm thickness fraction of 15-30% during the first three days of mechanical ventilation was associated with the shortest duration of mechanical ventilation and this may potentially help guide the management of respiratory support.

On the other hand, the effect of under-assist breathing or allowing excessive respiratory effort could be harmful. Some reported in chronic obstructive pulmonary disease (COPD) exacerbation patients found that the increased negative intra-thoracic pressure potentially causes injury to the diaphragm sarcomeres, which are the muscle fibers responsible for generating force during breathing and it was proportional to the degree of obstruction. And compared light microscopy of the diaphragmatic muscles necropsy in patients who died of COPD with normal subjects. They found muscular necrosis and accumulation of fibrosis and collagen deposits. The cytoplasm was scattered, disrupted, and lipofuscin accumulation with hyper-eosinophilia was observed.

In addition, an excessive high respiratory effort can cause lung injury by patient-self known as patient self-inflicted lung injury (P-SILI), a theory first mentioned that the increased magnitude of negative intrathoracic pressure during inhalation may cause the fluid shift from the pulmonary capillaries to the alveoli causing pulmonary edema. This is relevant to the observational studies that the occurrence of negative intrathoracic pressure during large inhalations in obstruction airway patients, such as tracheal stenosis, also results in pulmonary edema. In latterly confirmed this hypothesis. Subsequent studies have supported this phenomenon and overall could be explained through the increase of transpulmonary pressure, pendelluft phenomenon and patient-ventilator asynchrony (PVA).

However, no current studies determine the relationship between respiratory effort measurement during mechanical ventilation and clinical outcomes. Therefore, we conduct the study to determine the relationship between respiratory effort parameters and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged between 18-75 years.
2. Admitted to the critical care and semi-critical care units (ICUs) of the Department of -Internal Medicine, Ramathibodi Hospital (ICUs 9IC, 8IK, and 7NW).
3. Patients with acute respiratory failure admitted to the hospital with the following conditions within the first 48 hours:

   * PaO2/FiO2 greater than 150 or
   * PaO2 less than 60 mm Hg or
   * SaO2 less than 90 mm Hg or
   * Work of breathing more than 25 breaths per minute or requiring respiratory muscle assistance
4. Permission obtained from the attending physician.
5. Research participants or their direct relatives must sign informed consent.
6. The research can commence and data can be recorded within 48 hours after the patient has received treatment with the mechanical ventilator.

Exclusion Criteria:

1. Admitted to the hospital or had a history of hospital admission within a month before recruitment.
2. History of cardiovascular or cerebrovascular events within the last 12 months.
3. Pregnant.
4. Terminal-stage cancer patient, terminal illness-stage of disease who desire palliative care.
5. Active neurological or muscular disorders affecting stability.
6. Brain coma, brain death, or status epilepticus.
7. Severe mental health conditions, including active depression with psychotic features, bipolar disorder, or schizophrenia.
8. Uncontrolled thyroid conditions within a month before recruitment.
9. Uncorrectable patients with severe hypoxemia (P/F ratio less than 150).
10. Patients receiving neuromuscular blocking agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A single-center analytical observational prospective study was conducted between June 2022 and April 2024. We enrolled acute respiratory failure patients who required mechanical ventilation from the intensive care units (ICUs) at Ramathibodi Hospital, Mahidol University.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
28 days ventilator-free days (VFDs) | After intubated patients were recruited until successful extubation or dead/failed extubation with in 28 days.
  The number of VFDs was defined as the number of days from the last day of mechanical ventilation to day 28. If a patient died during the first 28 days, their number of VFDs is equal to zero.

SECONDARY OUTCOMES:
28 days all-cause mortality | After intubated patients were recruited until alive or dead with in 28 days.
  Short-term mortality was defined as death occurring within 28 days from the start of enrollment, documented as either alive or deceased 28 days after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Phruet Soipetkasem, Critical care doctor, Principal Investigator — Doctor of Critical care medicine Ramathibodi hospital; Pongdhep Theerawit, Assoc. Prof., Study Chair — Head of Critical care medicine Ramathibodi hospital; Yuda Sutherasan, Assoc. Prof., Study Director — Clinical professor of Pulmonary and Critical care medicine Ramathibodi hospital; Mr. Detajin Junhasavasdikul, Asst.Prof., Study Director — Clinical professor of Pulmonary and Critical care medicine Ramathibodi hospital
Locations (1):
- Mr. Phruet Soipetkasem, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Orozco-Levi M, Lloreta J, Minguella J, Serrano S, Broquetas JM, Gea J. Injury of the human diaphragm associated with exertion and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1734-9. doi: 10.1164/ajrccm.164.9.2011150. PMID 11719318
- [Background] Scott A, Wang X, Road JD, Reid WD. Increased injury and intramuscular collagen of the diaphragm in COPD: autopsy observations. Eur Respir J. 2006 Jan;27(1):51-9. doi: 10.1183/09031936.06.00143004. PMID 16387935
- [Background] Loeb L. The Mechanism in the Development of Pulmonary Edema. Proceedings of the Society for Experimental Biology and Medicine. 1928;25(5):321-323. doi:10.3181/00379727-25-3837
- [Background] Moore RL, Binger CA. THE RESPONSE TO RESPIRATORY RESISTANCE : A COMPARISON OF THE EFFECTS PRODUCED BY PARTIAL OBSTRUCTION IN THE INSPIRATORY AND EXPIRATORY PHASES OF RESPIRATION. J Exp Med. 1927 May 31;45(6):1065-80. doi: 10.1084/jem.45.6.1065. PMID 19869306
- [Background] Barach AL, Eckman M. THE EFFECTS OF INHALATION OF HELIUM MIXED WITH OXYGEN ON THE MECHANICS OF RESPIRATION. J Clin Invest. 1936 Jan;15(1):47-61. doi: 10.1172/JCI100758. No abstract available. PMID 16694380
- [Background] Dreyfuss D, Soler P, Basset G, Saumon G. High inflation pressure pulmonary edema. Respective effects of high airway pressure, high tidal volume, and positive end-expiratory pressure. Am Rev Respir Dis. 1988 May;137(5):1159-64. doi: 10.1164/ajrccm/137.5.1159. PMID 3057957
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Result] Mascheroni D, Kolobow T, Fumagalli R, Moretti MP, Chen V, Buckhold D. Acute respiratory failure following pharmacologically induced hyperventilation: an experimental animal study. Intensive Care Med. 1988;15(1):8-14. doi: 10.1007/BF00255628. PMID 3230208
- [Result] Yoshida T, Torsani V, Gomes S, De Santis RR, Beraldo MA, Costa EL, Tucci MR, Zin WA, Kavanagh BP, Amato MB. Spontaneous effort causes occult pendelluft during mechanical ventilation. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1420-7. doi: 10.1164/rccm.201303-0539OC. PMID 24199628
- [Result] Dzierba AL, Khalil AM, Derry KL, Madahar P, Beitler JR. Discordance Between Respiratory Drive and Sedation Depth in Critically Ill Patients Receiving Mechanical Ventilation. Crit Care Med. 2021 Dec 1;49(12):2090-2101. doi: 10.1097/CCM.0000000000005113. PMID 34115638
- [Result] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Result] Loring SH, O'Donnell CR, Behazin N, Malhotra A, Sarge T, Ritz R, Novack V, Talmor D. Esophageal pressures in acute lung injury: do they represent artifact or useful information about transpulmonary pressure, chest wall mechanics, and lung stress? J Appl Physiol (1985). 2010 Mar;108(3):515-22. doi: 10.1152/japplphysiol.00835.2009. Epub 2009 Dec 17. PMID 20019160
- [Result] Baedorf Kassis E, Loring SH, Talmor D. Mortality and pulmonary mechanics in relation to respiratory system and transpulmonary driving pressures in ARDS. Intensive Care Med. 2016 Aug;42(8):1206-13. doi: 10.1007/s00134-016-4403-7. Epub 2016 Jun 18. PMID 27318943
- [Result] Taran Z, Namadian M, Faghihzadeh S, Naghibi T. The Effect of Sedation Protocol Using Richmond Agitation-Sedation Scale (RASS) on Some Clinical Outcomes of Mechanically Ventilated Patients in Intensive Care Units: a Randomized Clinical Trial. J Caring Sci. 2019 Dec 1;8(4):199-206. doi: 10.15171/jcs.2019.028. eCollection 2019 Dec. PMID 31915621

DOCUMENTS (1):
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT06433076/ICF_000.pdf